CLINICAL TRIAL: NCT03175016
Title: Irinotecan-Eluting Bead (DEBIRI) for Unresectable Liver Metastases From Colorectal Cancer After Systemic Chemotherapy Failure
Brief Title: Irinotecan-Eluting Bead (DEBIRI) for Patients With Liver Metastases From Colorectal Cancer
Acronym: DEBIRI-CRLM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-CIH-IR-006
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Colon Cancer Liver Metastasis
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEBIRI (Experimental): Transcatheter arterial chemoembolization(TACE) with Irinotecan eluting-bead(DEBIRI)
  Interventions: Procedure: TACE; Drug: Irinotecan; Device: eluting-bead

INTERVENTIONS:
Procedure: TACE — Transcatheter arterial chemoembolization（TACE）is a minimally invasive procedure performed to restrict a tumor's blood supply.
  Other Names: Transcatheter arterial chemoembolization
Drug: Irinotecan — Irinotecan hydrochloride is a semisynthetic derivative of camptothecin, an alkaloid extracted from the tree Camptotheca acuminata. Irinotecan hydrochloride trihydrate is a pale yellow to yellow crystalline powder, it is mixed in eluting-beads and injected in the tumor.
Device: eluting-bead — The eluting-bead,loaded with irinotecan (DEBIRI) to treat patients with hepatic metastases from colorectal cancer.

SUMMARY:
This is a multicentre, open labeled, single arm study to determine effectiveness and safety of chemoembolization with Irinotecan-Eluting Bead(DEBIRI) in the treatment of unresectable liver metastases in patients with colorectal cancer after chemotherapy failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age, of any race or sex, who have histologic or radiologic proof of colorectal cancer to the liver, who are able to give informed consent, will be eligible.
2. Patients with primary colorectal lesions removed, and negative extrahepatic metastasis
3. Patients with at least one measurable liver metastases, with size > 2cm or less than 5 liver metastases,with size smaller than 10cm.
4. Patients have received at least six cycle system chemotherapy based irinotecan or oxaliplatin and got a failure outcome; or patients who are intolerance of operation.
5. No intervention therapy was received for liver lesions during one year.
6. Life expectancy of > 3 months
7. Child-pugh's grade A or B (no more than 7 score).
8. Eastern Cooperative Oncology Group (ECOG) Performance Status score of < 2
9. Signed, written informed consent

Exclusion Criteria:

1. Patients with extrahepatic metastasis
2. Patients has received TACE,ablation and iodine seed implantation for liver lesions during one year.
3. With obvious arterio-venous fistula
4. Patients suffered with other cancer(Except for cured basal or squamous cell skin cancer or cervical carcinoma in situ)
5. Hematologic function: leukocytes <3000cell/mm3, platelets<50000/mm3, with no hypersplenism.
6. Adequate renal function (creatinine ≤ 2.0mg/dl)
7. Alanine transaminase(ALT) and/or glutamic oxalacetic transaminase(AST) >5 times upper limit of normal(ULN)
8. International Normalized Ratio (INR) >1.5, or being treated by anticoagulants, or being suffered hemorrhagic disease.
9. With serious heart, kidney, bone marrow, or lung, central nervous system diseases.
10. With recent infections and received antibiotics.
11. Other conditions place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Tumor Response of two months | Two months post first treatment
  Response rate(RR)
Tumor Response of four months | four months post first treatment
  Response rate(RR)
Tumor Response of six months | Six months post first treatment
  Response rate(RR)

SECONDARY OUTCOMES:
overall survival | From date of first treatment until the date of death from any cause, whichever came first, assessed up to 24 months
  overall survival(OS)
Time to intrahepatic progression | From date of first treatment until the date of intrahepatic progression, whichever came first, assessed up to 24 months
  Time to intrahepatic progression(THP)
Time to extrahepatic progression | From date of first treatment until the date of extrahepatic progression, whichever came first, assessed up to 24 months
  Time to extrahepatic progression(TEP)
Quality of life | Six months post first treatment
  Assesment Quality of life by EORTC QOL-C30 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No